### University of California, Los Angeles

### RESEARCH INFORMATION SHEET

Targeted Upstream Prevention (T-UP) study

### INTRODUCTION

Lauren Wisk, PhD from the Division of General Internal Medicine in the Department of Medicine at the University of California, Los Angeles is conducting a research study. This study is being funded by the American Diabetes Association. You were selected as a possible participant in this study because you are currently enrolled (either full time or part time) as an undergraduate at UCLA and meet criteria for the T-UP Wellness Program, specifically reporting the presence of risk factors for cardiometabolic disease (e.g., type 2 diabetes) as outlined by the Centers for Disease Control and Prevention (CDC).

### WHAT SHOULD I KNOW ABOUT A RESEARCH STUDY?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

### WHY IS THIS RESEARCH BEING DONE?

The purpose of this research study is to test out a student-focused wellness program, based on the UC Diabetes Prevention Program, for feasibility, acceptability and impact on health and wellness outcomes, including risk factors for later cardiometabolic disease.

### HOW LONG WILL THE RESEARCH LAST AND WHAT WILL I NEED TO DO?

If you volunteer to participate in this study,

- You will be randomized to the order in which you receive program components. Some participants will receive the nutrition/exercise/stress program first and other participants will receive the substance use/financial literacy/study skills program first. Participants will then switch programs in the second academic year.
- Depending on which program you are randomized to receive first, you will be asked to complete the program either in-person, on-campus (including the Wooden Center, UCLA Teaching Kitchen) or virtually (via Zoom). For the in-person program, you will be asked to attend up to 18 in-person sessions, ranging from 60-75 minutes, no more than one session per week during the academic year (Fall, Winter, Spring quarters). For the remote program, you will be asked to attend a Zoom session to go over materials related to study habits (Fall quarter), alcohol use (Winter quarter), and financial literacy (Spring quarter). Zoom session is approximately 60 minutes.

- There are two assessments per year, baseline and 9-month follow-up for the first year and baseline and 9-month follow-up for the second year. These assessments will be done in October and June, respectively.
- We will ask you to complete two 30-minute surveys (baseline and 9-month follow-up) that asks questions about sociodemographics (e.g., age, sex, race, ethnicity, socioeconomic status), social vulnerability, health-related quality of life, mental health, self-perceived weight status and self-reported physical activity and diet. Surveys will be administered online.
- A research assistant will collect your height and weight measurements at baseline and 9-month follow-up. RA will meet you at the Wooden Center to collect your measurements.
- Participants will be asked to self-report weight at the end of the fall and winter quarter as intermediate check-ins; data will be collected via brief REDCap survey.
- In-person program participants will participate in a "Steps" challenge during the Fall, Winter, and Spring in-person sessions. Participants will be put into teams for this challenge.

### ARE THERE ANY RISKS IF I PARTICIPATE?

- Risks may include feeling uncomfortable with taking up your time.
- There may also be a risk of people learning that you participated in the study.
- In order to minimize these risks, you may withdraw your participation at any time.

### ARE THERE ANY BENEFITS IF I PARTICIPATE?

Free access to the wellness program.

### WHAT OTHER CHOICES DO I HAVE IF I CHOOSE NOT TO PARTICIPATE?

Your alternative to participating in this research study is to not participate.

## HOW WILL INFORMATION ABOUT ME AND MY PARTICIPATION BE KEPT CONFIDENTIAL?

The researchers will do their best to make sure that your private information is kept confidential. Information about you will be handled as confidentially as possible, but participating in research may involve a loss of privacy and the potential for a breach in confidentiality. Study data will be physically and electronically secured. As with any use of electronic means to store data, there is a risk of breach of data security.

## USE OF PERSONAL INFORMATION THAT CAN IDENTIFY YOU:

All research data will be de-identified at the end of the study. We will provide our data resources on https://figshare.com/, a general data repository. De-identified data may be shared with other researchers upon application and reasonable request per funder requirements.

### How information about you will be stored:

Only the PI and a designated member of the research team will have access to personal information. All data (contact information, questionnaires and eligibility criteria data) will be stored on the PI's desktop computer in the PI's office, and backed up to a password-protected external hard drive. Information will also be stored in an encrypted and secure server. Only members of the research team will have access to the data.

## People and agencies that will have access to your information:

The research team will have access to study data and records to monitor the study. Research records provided to authorized, non-UCLA personnel will not contain identifiable information about you. Publications and/or presentations that result from this study will not identify you by name.

Employees of the University may have access to identifiable information as part of routine processing of your information, such as processing payment. However, University employees are bound by strict rules of confidentiality.

### WILL I BE PAID FOR MY PARTICIPATION?

Participants will be compensated with ≥\$100 for completing all study components. Participants will be compensated with a \$40 gift card after completion of the baseline survey, a \$60 gift card after completion of the 9-month follow survey, and a \$10 gift card after completion of 15 out of the 18 acceptability surveys (in-person program). Furthermore, all members of the winning team for the "Steps" challenge will receive a \$5 gift card. Lastly, we will provide a workout pass to inperson program participants. We will provide these vouchers for each quarter in which attendance in the prior quarter was at least 75% (e.g., if they attended 75% of the fall quarter sessions they will receive a free voucher for all winter quarter).

# WHO CAN I CONTACT IF I HAVE QUESTIONS ABOUT THIS PROGRAM? The research team:

If you have any questions, comments or concerns about the program, you can talk to one of the researchers. Please contact: Dr. Lauren Wisk (Principal Investigator) at 310-267-5308 or lwisk@mednet.ucla.edu; and/or, the research team at 310-592-3213 (call or text) or tupwellness@mednet.ucla.edu.

## **UCLA Office of the Human Research Protection Program (OHRPP):**

If you have questions about your rights as a participant, or you have concerns or suggestions and you want to talk to someone other than the researchers, you may contact the UCLA OHRPP by phone: (310) 206-2040; by email: participants@research.ucla.edu or by mail: Box 951406, Los Angeles, CA 90095-1406.

### WHAT ARE MY RIGHTS IF I TAKE PART IN THIS STUDY?

- You can choose whether or not you want to be in this study, and you may withdraw your consent and discontinue participation at any time.
- Whatever decision you make, there will be no penalty to you, and no loss of benefits to which you were otherwise entitled.

## USE OF DATA FOR FUTURE RESEARCH

Your data, including de-identified data may be kept for use in future research.